CLINICAL TRIAL: NCT07089537
Title: Acute Effects of Progressive Muscle Relaxation on Brain Waves, Heart Rate Variability, Muscle Tone, and Mental Stress
Brief Title: Acute Effects of Progressive Muscle Relaxation on Brain Waves
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kaohsiung Medical University (Other)
Responsible Party: Principal Investigator, Hsinyu Sun, graduate student, Kaohsiung Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: KMUHIRB-E(I)-20240388
Record Dates: First submitted 2025-03-13; First posted 2025-07-28 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Progressive Muscle Relaxation
MeSH Terms: interventions — RE1-silencing transcription factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- progressive muscle relaxation (Experimental): Participants will undergo approximately 30 minutes of Progressive Muscle Relaxation (PMR). Prior to the session, a brief introduction to the basic concepts of PMR will be provided. Participants will be instructed to close their eyes and focus on the sensations in their muscles. Following verbal instructions, they will sequentially contract and relax 14 major muscle groups from top to bottom. For each muscle group, participants will be asked to contract the muscles as strongly as possible for 7 seconds, followed by a 45-second relaxation period. This process will be repeated twice for each muscle group.
  Interventions: Other: progressive muscle relaxaiton; Other: Rest
- rest (Placebo Comparator): rest in a semi-recumbent position with eyes closed for 30 minutes, without any additional intervention.
  Interventions: Other: progressive muscle relaxaiton; Other: Rest

INTERVENTIONS:
Other: progressive muscle relaxaiton — Participants will undergo approximately 30 minutes of Progressive Muscle Relaxation (PMR). Prior to the session, a brief introduction to the basic concepts of PMR will be provided. Participants will be instructed to close their eyes and focus on the sensations in their muscles. Following verbal instructions, they will sequentially contract and relax 14 major muscle groups from top to bottom. For each muscle group, participants will be asked to contract the muscles as strongly as possible for 7 seconds, followed by a 45-second relaxation period. This process will be repeated twice for each muscle group.
Other: Rest — Rest in a semi-recumbent position with eyes closed for 30 minutes, without any additional intervention.

SUMMARY:
In modern environments, stress is present regardless of age or social role. Stress does not always have negative effects; in fact, it is a necessary response for survival, known as the stress response. This response includes increased heart rate, blood pressure, blood glucose levels, and decreased alpha brainwave activity. These physiological changes are primarily regulated by the sympathetic and parasympathetic branches of the autonomic nervous system, enabling us to cope with environmental threats. However, when the stress response system becomes overwhelmed or imbalanced-whether due to accumulated chronic stress or acute stress-it may result in adverse effects on both physical and mental health.

Relaxation techniques are non-pharmacological methods that promote parasympathetic nervous system activity. The goal is to reduce excessive arousal, alleviate anxiety, slow down thought processes, and relieve stress, thereby achieving relaxation in a natural way. These methods help lower blood pressure, improve circulation, relax muscles, and enhance concentration. Previous studies have demonstrated a correlation between relaxation and attention, suggesting that relaxation can improve attentional efficiency. Moreover, it is well-documented that executive function tends to decline under stress. Relaxation techniques are commonly incorporated into psychological therapies, yet they are more accessible, easier to practice, and can be conveniently performed at home.

Therefore, the aim of this study is to investigate whether PMR can produce immediate relaxation effects as measured by EEG (cortical excitability), heart rate variability, and muscle tone, and whether it can improve performance under psychological stress. The goal is to further explore the potential application of PMR in healthy populations facing acute stress conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* Age: 18 years and above
* Body Mass Index (BMI) between 18 and 24
* Able to remain in a semi-recumbent position for 2 hours

Exclusion Criteria:

* Individuals with communication impairments or difficulty understanding instructions
* Color vision deficiency
* Open wounds or injuries on the scalp
* Currently taking medications that affect cardiovascular or autonomic nervous system regulation
* Muscle strain or pain

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2025-02-24 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Electroencephalography | 20 min in total
  Analysis of changes in EEG band power excitability across the frontal, central, and occipital brain regions.

SECONDARY OUTCOMES:
Muscle tension | 15 mins
  Changes in muscle tension
heart rate variability | 20 mins in total
  changes in frequency domain heart rate variability
Self-Assessment Manikin | 1min
  Whether the subjective emotion is calm or excited

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Medical University, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No